CLINICAL TRIAL: NCT02742389
Title: A Telephone Call to Decrease Patient Anxiety Before Urodynamic Testing: a Randomized Controlled Trial
Brief Title: Urodynamic Testing: Can we Improve Patient Experience?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Urogynecology Associates (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Lekha S. Hota, MD, Boston Urogynecology Associates
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 004-2016
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Urinary Incontinence; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard counseling (No Intervention): This group will receive the standard counseling that all our patients would receive if they are scheduled to have urodynamic testing. This counseling will include a description of the procedure and a handout about urodynamic testing
- Standard + Preprocedure Telephone Call (Other): The participants will receive the standard counseling that all our patients who are scheduled for urodynamic testing receive (just like those who are assigned to group 1). In addition, the participants will receive intervention: a pre-procedural telephone call from the investigators 1 week before their testing to talk about the procedure.
  Interventions: Other: Preprocedure Telephone Call

INTERVENTIONS:
Other: Preprocedure Telephone Call — The participants will receive a phone call from the investigators 1 week before their testing to talk about the procedure and answer any questions that patients may have . The investigator calling the participant will document the duration of the phone call and any questions asked by the participant
  Arms: Standard + Preprocedure Telephone Call

SUMMARY:
The purpose of this study is to determine whether an intervention (pre-procedure telephone call by the investigators) will reduce anxiety in women undergoing urodynamic testing (UDT) compared to usual care. Our hypothesis is that women who receive the intervention will report less anxiety immediately before UDT than women who receive usual care.

DETAILED DESCRIPTION:
This is a non-blinded, randomized controlled trial. The clinical trial will investigate whether a telephone call by the investigator one week prior to urodynamic testing (UDT) will decrease patient pre-procedure anxiety, improve patient-reported preparedness and increase satisfaction compared to usual care. Patients who are scheduled for UDT will be informed about the study. If the patient agrees to participate in the study, she will be randomized to one of 2 groups based on the week of her scheduled UDT.

Group 1: Standard counseling. This group will receive the standard counseling that all Boston Urogynecology Associates (BUA) patients would receive if they are scheduled to have urodynamic testing. This counseling will include a description of the procedure and a handout about urodynamic testing. On the day of their test the participants will be asked to complete a brief survey about their experience before and after their testing. The investigators will also collect some information from their medical record, such as age and prior urogynecologic procedures.

Group 2: Standard counseling plus the intervention. The participants assigned to be in the intervention group will receive the standard counseling that all BUA patients who are scheduled for urodynamic testing receive (just like those who are assigned to group 1). This counseling includes a description of the procedure and a handout about urodynamic testing. In addition, the participants will receive a phone call from the investigators 1 week before their testing to talk about the procedure. The investigator calling the participant will document the duration of the phone call and any questions asked by the participant. On the day of their test the participants will be asked to complete the same surveys as group 1.

Surveys given to the participants on the day of their UDT appointment will include:

1. A pre-UDT questionnaire that includes questions on demographics, overall anxiety, anxiety about specific elements of procedure, self-reported preparedness and satisfaction.
2. A brief post-UDT questionnaire addressing test experience and pain.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or greater
2. Female
3. Patients who have decided to schedule Urodynamic Testing to follow-up lower urinary tract dysfunction, pelvic organ prolapse, and/or urinary incontinence

Exclusion Criteria:

1. Pregnant
2. Presence of indwelling catheters
3. History of prior Urodynamic Testing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Overall pre-procedure anxiety as measured on a visual analog scale. | Day 1
  Overall pre-procedure anxiety as measured on a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lekha Hota, MD, Principal Investigator — Mount Auburn Hospital
Locations (1):
- Mount Auburn Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No